CLINICAL TRIAL: NCT05759702
Title: Correlation Between Body Mass Index, Manual Dexterity and Handgrip Strength in School Aged Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Wessam Osama Sayed, demonstrator, Cairo University
Other Study IDs: P.T.REC/012/004242
Record Dates: First submitted 2023-02-26; First posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Body Mass Index,Manual Dexterity,Handgrip Strength,School Aged Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- normal weight: normal weight students will be enrolled in this group their BMI range from 5th percentile to less than the 85th percentile on CDC growth chart
- overweight: overweight students will be enrolled in this group their BMI range from 85th to less than the 95th percentile on CDC growth chart
- obese: obese students will be enrolled in this group their BMI range from Equal to or greater than the 95th percentile on CDC growth chart

SUMMARY:
The purpose of current study is to investigate the relation between body mass index, manual dexterity and handgrip strength in school aged children having normal weight, overweight and obesity.

DETAILED DESCRIPTION:
The study targeted the normal weight, overweight and obese students (9-11) from both sexes will be selected from governmental primary schools.

Study design:

Cross sectional observational correlational study.

A. Inclusion criteria:

1. The students' age ranges from 9 to 11 years.
2. Normal weight, Overweight and obese students were included
3. both boys and girl will be included.

B. Exclusion criteria:

The students will be excluded from the study if they have one of the following:

1. Congenital abnormalities or medical conditions, which may affect the study.
2. Musculoskeletal problems such as previous or recent orthopedic surgery, fractures, prostheses, inflammation of the fingers, arms, or shoulder.
3. Visual or hearing defects.
4. Motor, behavioral, or neurologic disorders and learning disabilities.

   * All children will be assessed using: the Standard weight and height measuring scale to determine their BMI.
   * Assessment of manual dexterity will be carried out by using the Bruininks-Oseretsky Test of Motor Proficiency, Second Edition (BOT-2) (Bruininks and Bruininks, 2005).
   * Handgrip strength will be assessed by hand dynamometer.

ELIGIBILITY:
Inclusion Criteria:

1. The students' age will range from 9 to 11 years.
2. Normal weight, Overweight and obese students including both boys and girl.

Exclusion Criteria:

* The students will be excluded from the study if they have one of the following:

  1. Congenital abnormalities or medical conditions, which may affect the study.
  2. Musculoskeletal problems such as previous or recent orthopedic surgery, fractures, prostheses, inflammation of the fingers, arms, or shoulder.
  3. Visual or hearing defects.
  4. Motor, behavioral, or neurologic disorders and learning disabilities.

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
assessment of manual dexterity | Baseline-45min for each participant
  assessment of manual dexterity will be carried out by using using the Bruininks-Oseretsky Test of Motor Proficiency, Second Edition (BOT-2) (Bruininks and Bruininks, 2005).
• Handgrip strength | Baseline-45min for each participant
  • Handgrip strength will be assessed by hand dynamometer device

CONTACTS AND LOCATIONS:
Overall Officials: wessam os sayed, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt